CLINICAL TRIAL: NCT04609618
Title: A Prospective, Self-controlled, Feasibility Study to Evaluate Appscent Device Safety and Effectiveness for Relief of Obstructive Sleep Apnea (OSA) Syndrome in Adults.
Brief Title: Evaluatation of Appscent Device Safety and Effectiveness for Relief of Obstructive Sleep Apnea (OSA) Syndrome in Adults.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Y.A. Appscent Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN001
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Prospective, self-controlled, feasibility study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obstructive Sleep Apnea patients (Experimental): Appscent device will discharge odor during the in lab night sleep
  Interventions: Device: Appscent Device

INTERVENTIONS:
Device: Appscent Device — computer-controlled, low pressure compressed air based, with disposable odorant capsules solution provided an odor environment at the nose,

SUMMARY:
Obstructive Sleep Apnea (OSA) syndrome is a disorder characterized by repetitive episodes of upper airway obstruction that occur during sleep.

The standard treatment for apnea remains a device consisting of a pump and nasal mask that provide continuous positive airway pressure (CPAP). The major disadvantage of CPAP is the relatively low compliance.

Appscent developed a non-contact effortless bedside solution based on the following: odors modify respiratory patterns during wake . Mildly trigeminal and pure olfactory odorants do not arouse or wake.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) syndrome is a disorder characterized by repetitive episodes of upper airway obstruction that occur during sleep. OSA lead to desaturation and often lead to an arousal.

Associated features include loud snoring and fragmented non-refreshing sleep and have profound impact on quality of life, on safety on the roads and at work, and on the cardiovascular and metabolic systems.

The standard treatment for apnea remains a device consisting of a pump and nasal mask that provide continuous positive airway pressure (CPAP). CPAP acts as a pneumatic splint that elevates and maintains a constant pressure along the upper airway during inspiration and expiration that prevents airway collapse. The major disadvantage of CPAP is the relatively low compliance.

Appscent developed a non-contact effortless bedside solution based on the following: odors modify respiratory patterns during wake . Mildly trigeminal and pure olfactory odorants do not arouse or wake. Odorants transiently presented during sleep induced a respiratory rejection type response, this suggests that manipulating the respiratory system without waking is viable .

ELIGIBILITY:
Inclusion Criteria:

1. OSA diagnosed; AHI≥20
2. Male and Female Aged 40 to 70 years old
3. Patients of childbearing potential must agree to use methods of contraception and have negative pregnancy test at screening. Effective methods of contraception must be used throughout the study
4. BMI< 35
5. Patient is willing and able to give his/her written informed consent

Exclusion Criteria:

1. Chronic lung disease (including Asthma and COPD)
2. Congestive Heart Failure
3. Exhibiting any flu-like or upper respiratory illness symptoms at time of assessment
4. History of severe nasal allergies or sinusitis or difficulty breathing through the nose
5. Persistent blockage of one or both nostrils
6. Any previous operation or trauma to the nose
7. Previous diagnosis of insomnia, narcolepsy, periodic limb movement disorder, respiratory failure
8. Any use of antipsychotic, Hypnotic drugs
9. Major neurological diagnosis
10. Active malignant disease including chemotherapy or radiotherapy treatment
11. Pregnant or lactating women
12. Drug abuse
13. Medical history of epilepsy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Safety event frequency | 3 weeks
  Device or treatment-related adverse events.

SECONDARY OUTCOMES:
Sleepiness effect | 2 weeks
  Overall sleepiness change measured by ESS

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Lab, Tel Aviv, Israel